CLINICAL TRIAL: NCT05663073
Title: A Randomized, Open-label, Crossover, Phase 1 Study to Evaluate Pharmacokinetics and Safety of Irbesartan/Amlodipine Fixed Dose Combination in Comparison With Co-administration of Mono Compounds in Healthy Volunteers
Brief Title: Pharmacokinetics of Irbesartan/Amlodipine FDC and Co-administration of Irbesartan and Amlodipine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HD-AI-101
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irbesartan/Amlodipine Fixed dose combination (Experimental): participants will receive one tablet of Irbesartan/Amlodipine FDC in a crossover design
  Interventions: Drug: Irbesartan/Amlodipine FDC
- Co-administration of Irbesartan and Amlodipine (Experimental): participants will receive one table each of Irbesartan and Amlodipine in a crossover design
  Interventions: Drug: Irbesartan; Drug: Amlodipine

INTERVENTIONS:
Drug: Irbesartan/Amlodipine FDC — Irbesartan/Amlodipine FDC
  Arms: Irbesartan/Amlodipine Fixed dose combination
Drug: Irbesartan — Co-administration of Irbesartan and Amlodipine
  Arms: Co-administration of Irbesartan and Amlodipine
Drug: Amlodipine — Co-administration of Irbesartan and Amlodipine
  Arms: Co-administration of Irbesartan and Amlodipine

SUMMARY:
The purpose of this study is to compare pharmacokinetics and safety of Irbesartan and Amlodipine Fixed Dose Combination and coadministration of mono compounds in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older on screening
* Signed informed consent
* Healthy Volunteer
* Other inclusion applies

Exclusion Criteria:

* Clinically relevant/significant findings as evaluated by the investigator
* Other exclusion applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
AUCt of Irbesartan and Amlodipne | 72 hours
Cmax of Irbesartan and Amlodipne | 72 hours

SECONDARY OUTCOMES:
AUCinf of Irbesartan and Amlodipine | 72 hours
AUCt/AUCinf of Irbesartan and Amlodipine | 72 hours
tmax of Irbesartan and Amlodipine | 72 hours
half-life of Irbesartan and Amlodipine | 72 hours
CL/F of Irbesartan and Amlodipine | 72 hours
Vz/F of Irbesartan and Amlodipine | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea